CLINICAL TRIAL: NCT04489784
Title: Effects of the Infrared Laser on Classical Ballerinas' Feet
Brief Title: Infrared Laser and Classical Ballerinas' Feet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fernanda Rossi Paolillo, Professor, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ballet
Record Dates: First submitted 2020-07-20; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Pain
Keywords: Pain; Feet; Ballerinas
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: To evaluate the immediate and long-term effects of infrared laser on classical ballerinas' feet.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Laser treatment on ballerina's feet.
  Interventions: Device: Infrared Laser

INTERVENTIONS:
Device: Infrared Laser — An aluminum gallium arsenide (AlGaAs) diode laser device (Twin laser, MMOptics, São Carlos, SP, Brazil) was used. The irradiation parameters were as follows: infrared laser (808 nm wavelength) with a spot area of 0.04 cm2, and an average optical power of 100 mW operated in a continuous mode during 1 minute per point, leading to an irradiance of 2,500 mW/cm2, energy of 6 J and fluence of 125 J/cm2 per point. The laser was applied on ballerina's feet twice a week during three months.

SUMMARY:
Overuse injuries and painful symptoms in athletes and dancers (especially classical ballerinas) may lead to reduced functional performance. However, laser application may reduce pain and increase physical conditioning. The aim of the current study was to evaluate the immediate and long-term effects of infrared laser on classical ballerinas' feet. The hypothesis investigators was that the infrared laser would be able to reduce pain perception and enhance functional performance in ballerinas.

DETAILED DESCRIPTION:
High risk of injuries and painful symptoms in athletes and dancers (especially classical ballerinas) may lead to reduced functional performance. The use of photobiomodulation may improve functional performance in ballerinas that are affected by foot pain. An aluminum gallium arsenide (AlGaAs) diode laser device was uded. Infrared laser (808 nm) was applied on ballerina's feet twice a week during three months. Thermography, algometry and unipodal static standing balance test were performed. There were pain relief and improvement of functional performance in ballerinas.

ELIGIBILITY:
Inclusion Criteria:

- Female adults who perform classical ballet training and feel pain in their foot

Exclusion Criteria:

- The occurrence of injuries in the last 6 months

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Analysis of pain for feet by algometry | 3 months
  Pressure pain thresholds (PPT) were assessed with an electronic algometer. The pressure was applied and the ballerinas were instructed to ask to say "stop" when the sensation changed from pressure to pain. Three PPT measurements were performed to obtain an average.
Analysis of pain for feet by the visual analogue pain intensity scale | 3 months
  A continuous scale comprised of a horizontal line with 10 centimeters in length was used. All ballerinas were instructed to make a mark with a pen at any point on the line between 2 verbal descriptors, one for each symptom extreme ["No pain" (score=0) and "as bad as it could be" or "worst imaginable pain" (score=10)].

SECONDARY OUTCOMES:
Balance Test | 3 months
  Static Standing Balance Test was performed. Ballerinas were instructed to stand on one foot to a maximum of one minute. The time was measured in seconds.
Thermal Analysis | 3 months
  Cutaneous temperatures of ballerina's feet were analyzed by thermography.

CONTACTS AND LOCATIONS:
Locations (1):
- Fernanda Rossi Paolillo, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Leal Junior EC, Lopes-Martins RA, Rossi RP, De Marchi T, Baroni BM, de Godoi V, Marcos RL, Ramos L, Bjordal JM. Effect of cluster multi-diode light emitting diode therapy (LEDT) on exercise-induced skeletal muscle fatigue and skeletal muscle recovery in humans. Lasers Surg Med. 2009 Oct;41(8):572-7. doi: 10.1002/lsm.20810. PMID 19731300
- [Background] Paolillo FR, Paolillo AR, Joao JP, Frasca D, Duchene M, Joao HA, Bagnato VS. Ultrasound plus low-level laser therapy for knee osteoarthritis rehabilitation: a randomized, placebo-controlled trial. Rheumatol Int. 2018 May;38(5):785-793. doi: 10.1007/s00296-018-4000-x. Epub 2018 Feb 26. PMID 29480363
- [Background] Adabbo M, Paolillo FR, Bossini PS, Rodrigues NC, Bagnato VS, Parizotto NA. Effects of Low-Level Laser Therapy Applied Before Treadmill Training on Recovery of Injured Skeletal Muscle in Wistar Rats. Photomed Laser Surg. 2016 May;34(5):187-93. doi: 10.1089/pho.2015.4031. Epub 2016 Apr 8. PMID 27058781
- [Background] Shah S. Determining a young dancer's readiness for dancing on pointe. Curr Sports Med Rep. 2009 Nov-Dec;8(6):295-9. doi: 10.1249/JSR.0b013e3181c1ddf1. PMID 19904068